CLINICAL TRIAL: NCT03374930
Title: Influence of Oesophageal Contractile Reserve in High Resolution Manometry on Post Operative Dysphagia After Anti-reflux Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EREDYS
Record Dates: First submitted 2017-12-12; First posted 2017-12-15 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multiple rapid swallows test (Other): Multiple rapid swallows test consists in giving to patient 4 to 6 sips of 2 mL of water, with an interval less than 4 seconds between the different sips.
  Interventions: Procedure: Multiple rapid swallows test

INTERVENTIONS:
Procedure: Multiple rapid swallows test — Multiple rapid swallows test consists in giving to patient 4 to 6 sips of 2 mL of water, with an interval less than 4 seconds between the different sips.

SUMMARY:
The main objective of this study is to evaluate, in a prospective cohort, the link between preoperative contractile reserve of oesophagus evaluated by high resolution manometry (HRM) and the occurrence of post operative dysphagia after anti-reflux surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an indication validated at a fundoplication directed by a visceral surgeon from Vienne county
* Patient sent for the realization of a preoperative HRM,
* Patient giving consent to participate in the study.

Exclusion Criteria:

* Patient unable to sign a consent or protected (minors, pregnant women, patient under guardianship),
* History of oesophageal surgery or radiotherapy,
* History of systemic pathology with oesophageal involvement,
* Contraindication to an oesophageal manometry : altered general status and vigilance , important swallowing disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2021-06-12 (Actual); Study Completion 2021-06-12 (Actual)

PRIMARY OUTCOMES:
presence of dysphagia | 3 months
  clinically evaluated by the surgeon

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Center, Poitiers, France

IPD SHARING:
Plan to Share IPD: No